CLINICAL TRIAL: NCT06298032
Title: A Placebo-controlled, Within-group Randomised, and Double-blind Trial Investigating Safety, Tolerability, and Pharmacokinetics of FE 999301 After Ascending Single and Multiple Doses in Healthy Subjects
Brief Title: A Study Investigating the Safety, Tolerability, Immunogenicity and Pharmacokinetics of Olamkicept in Healthy Persons
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000414
Record Dates: First submitted 2024-02-01; First posted 2024-03-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Olamkicept - Part A (Experimental)
  Interventions: Drug: Olamkicept Part A
- Placebo - Part A (Placebo Comparator)
  Interventions: Drug: Placebo
- Olamkicept - Part B (Experimental)
  Interventions: Drug: Olamkicept Part B
- Placebo - Part B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olamkicept Part A — Intravenous infusion. Single dose.
  Part A consists of 3 different doses
  * 1200 mg
  * 1800 mg
  * 2400 mg
  Other Names: FE 999301
  Arms: Olamkicept - Part A
Drug: Olamkicept Part B — Intravenous infusion. Multiple doses.
  Part B consists of 3 different doses.
  * 1200 mg
  * 1800 mg
  * 2400 mg
  Other Names: FE 999301
  Arms: Olamkicept - Part B
Drug: Placebo — Intravenous infusion
  Arms: Placebo - Part A; Placebo - Part B

SUMMARY:
Interleukin (IL)-6 is a cytokine produced in response to infection and tissue damage. IL-6 is believed to act as a key mediator in chronic inflammation and autoimmune diseases such as inflammatory bowel diseases. IL-6 is known to be involved in at least two distinct signalling pathways, classical and trans-signalling. The hypothesis is that classical signalling by IL-6 infers some beneficial effects (e.g. on gut barrier function), while excessive IL-6 trans-signalling may have detrimental effects. Olamkicept (FE 999301) has been shown in vitro to be a selective IL-6 trans-signalling inhibitor, and administered at lower doses (600 mg every 2nd week for 12 weeks) it has proven to induce clinical improvement for patients with ulcerative colitis. The aim of this trial is to investigate safety, tolerability, immunogenicity and pharmacokinetics of Olamkicept at higher doses (up to 2400 mg) to support the clinical development program. Our hypothesis is that treatment with higher doses of Olamkicept will result in greater clinical improvement for patients with inflammatory bowel diseases.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥18 and ≤45 years of age at screening
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations, as assessed by the investigator (or designee) at screening and on Day -1

Exclusion Criteria:

* History of clinically significant medical conditions including, but not limited to, diseases of the renal, hepatic, respiratory, gastrointestinal, cardiovascular, neurological, musculoskeletal, psychiatric, immunological, haematological, oncological, endocrine, and metabolic systems and allergic diseases (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 49 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events, including type, intensity, and causality | End of trial (up to 64 days)
Change in vital signs from baseline to Day 36 after a single dose infusion | From baseline up to and including Day 36 after a single dose infusion
  Number of participants with clinically significant abnormal findings in vital signs (systolic blood pressure, diastolic blood pressure, pulse, body temperature), from baseline up to and including Day 36 after a single dose infusion (part A of the study).
Change in vital signs from baseline to Day 64 after multiple dose infusions | From baseline up to and including Day 64 after multiple dose infusions
  Number of participants with clinically significant abnormal findings in vital signs (systolic blood pressure, diastolic blood pressure, pulse, body temperature), from baseline up to and including Day 64 after multiple dose infusions (part B of the study)
Change in 12-lead electrocardiogram (ECG) from baseline to Day 36 after a single dose infusion | From baseline up to and including Day 36 after a single dose infusion
  Number of participants with clinically significant abnormal findings in ECG (heart rate, PR interval, RR, QRS duration, QT interval, QTc interval, QRS axis), from baseline up to and including Day 36 after a single dose infusion (part A of the study)
Change in 12-lead electrocardiogram (ECG) from baseline to Day 64 after multiple dose infusions | From baseline up to and including Day 64 after multiple dose infusions
  Number of participants with clinically significant abnormal findings in ECG (heart rate, PR interval, RR, QRS duration, QT interval, QTc interval, QRS axis), from baseline up to and including Day 64 after multiple dose infusions (part B of the study)
Change in haematology from baseline to Day 36 after a single dose infusion | From baseline to Day 36 after a single dose infusion
  Number of participants with clinically significant abnormal findings in haematology (haematocrit, haemoglobin, mean cellular volume (MCV), mean corpuscular haemoglobin content (MCH), mean corpuscular haemoglobin concentration (MCHC), platelet count, red blood cell count, reticulocytes, white blood cell count with differential count, neutrophils, eosinophils, basophils, lymphocytes, monocytes), from baseline up to and including Day 36 after a single dose infusion (part A of the study)
Change in haematology from baseline to Day 64 after multiple dose infusions | From baseline to Day 64 after multiple dose infusions
  Number of participants with clinically significant abnormal findings in haematology (haematocrit, haemoglobin, mean cellular volume (MCV), mean corpuscular haemoglobin content (MCH), mean corpuscular haemoglobin concentration (MCHC), platelet count, red blood cell count, reticulocytes, white blood cell count with differential count, neutrophils, eosinophils, basophils, lymphocytes, monocytes), from baseline up to and including Day 64 after multiple dose infusions (part B of the study)
Change in clinical chemistry from baseline to Day 36 after a single dose infusion | From baseline to Day 36 after a single dose infusion
  Number of participants with clinically significant abnormal findings in clinical chemistry (alanine aminotransferase (ALT), albumin, alkaline phosphatase, aspartate aminotransferase (AST), glucose, calcium, chloride, cholesterol, C-reactive protein, creatinine, estimated glomerular filtration rate (eGFR), gamma-glutamyltransferase, phosphate, potassium, sodium, thyroid stimulating hormone, free triiodothyronine, free thyroxine, total bilirubin, urea (blood urea nitrogen)), from baseline up to and including Day 36 after a single dose infusion (part A of the study)
Change in clinical chemistry from baseline to Day 64 after multiple dose infusions | From baseline up to and including Day 64 after multiple dose infusions
  Number of participants with clinically significant abnormal findings in clinical chemistry (alanine aminotransferase (ALT), albumin, alkaline phosphatase, aspartate aminotransferase (AST), glucose, calcium, chloride, cholesterol, C-reactive protein, creatinine, estimated glomerular filtration rate (eGFR), gamma-glutamyltransferase, phosphate, potassium, sodium, thyroid stimulating hormone, free triiodothyronine, free thyroxine, total bilirubin, urea (blood urea nitrogen)), from baseline up to and including Day 64 after multiple dose infusions (part B of the study)
Change in haemostasis parameters from baseline to Day 36 after a single dose infusion | From baseline up to and including Day 36 after a single dose infusion
  Number of participants with clinically significant abnormal findings in haemostasis parameters (activated partial thromboplastin time, prothrombin time) from baseline up to and including Day 36 after a single dose infusion (part A of the study)
Change in haemostasis parameters from baseline to Day 64 after multiple dose infusions | From baseline up to and including Day 64 after multiple dose infusions
  Number of participants with clinically significant abnormal findings in haemostasis parameters (activated partial thromboplastin time, prothrombin time) from baseline up to and including Day 64 after multiple dose infusions (part B of the study)
Change in urinalysis parameters from baseline to Day 36 after a single dose infusion | From baseline to Day 36 after a single dose infusion
  Number of participants with clinically significant abnormal findings in urinalysis parameters (protein, glucose, bilirubin, pH, nitrite, ketone, urobilinogen, blood, leukocytes, specific gravity) from baseline up to and including Day 36 after a single dose infusion (part A of the study)
Change in urinalysis parameters from baseline to Day 64 after multiple dose infusions | From baseline up to and including Day 64 after multiple dose infusions
  Number of participants with clinically significant abnormal findings in urinalysis parameters (protein, glucose, bilirubin, pH, nitrite, ketone, urobilinogen, blood, leukocytes, specific gravity) from baseline up to and including Day 64 after multiple dose infusions (part B of the study)

SECONDARY OUTCOMES:
Single-dose PK of FE 999301: Area under the concentration-time curve from dosing to infinity (AUCinf) | From baseline up to and including Day 36 after a single dose infusion
Single-dose PK of FE 999301: Area under the concentration-time curve to last measurable concentration (AUClast) | From baseline up to and including Day 36 after a single dose infusion
Single-dose PK of FE 999301: Observed plasma concentration at end of infusion (AUCeoi) | From baseline up to and including Day 36 after a single dose infusion
Single-dose PK of FE 999301: Baseline adjusted maximum observed concentration; also referred to as maximum exposure (Cmax) | From baseline up to and including Day 36 after a single dose infusion
Single-dose PK of FE 999301: Time of maximum observed concentration (tmax) | From baseline up to and including Day 36 after a single dose infusion
Single-dose PK of FE 999301: Terminal half-life (t1/2) | From baseline up to and including Day 36 after a single dose infusion
Single-dose PK of FE 999301: Mean residence time (MRT) | From baseline up to and including Day 36 after a single dose infusion
Single-dose PK of FE 999301: Total clearance (CL) | From baseline up to and including Day 36 after a single dose infusion
Single-dose PK of FE 999301: Apparent volume of distribution at steady-state (Vss) | From baseline up to and including Day 36 after a single dose infusion
Multiple-dose PK of FE 999301: Area under concentration-time curve from dosing up to time τ, where τ is the dosing interval (AUCτ) | From baseline up to and including Day 64 after a multiple dose infusions
Multiple-dose PK of FE 999301: Area under the concentration-time curve to last measurable concentration (AUClast) | From baseline up to and including Day 64 after a multiple dose infusions
Multiple-dose PK of FE 999301: Observed accumulation index (Rac) | From baseline up to and including Day 64 after a multiple dose infusions
Multiple-dose PK of FE 999301: Observed plasma concentration at end of infusion (Ceio) | From baseline up to and including Day 64 after a multiple dose infusions
Multiple-dose PK of FE 999301: Baseline adjusted maximum observed concentration; also referred to as maximum exposure (Cmax) | From baseline up to and including Day 64 after a multiple dose infusions
Multiple-dose PK of FE 999301: Time of maximum observed concentration (tmax) | From baseline up to and including Day 64 after a multiple dose infusions
Multiple-dose PK of FE 999301: Terminal half-life (t½) | From baseline up to and including Day 64 after a multiple dose infusions
Multiple-dose PK of FE 999301: Mean residence time (MRT) | From baseline up to and including Day 64 after a multiple dose infusions
Multiple-dose PK of FE 999301: Total clearance (CL) | From baseline up to and including Day 64 after a multiple dose infusions
Multiple-dose PK of FE 999301: Apparent volume of distribution at steady-state (Vss) | Day 64
Presence of anti-FE 999301 antibodies on Days 1, 15, and 57 after multiple dose infusions | On Days 1, 15, and 57 after multiple dose infusions

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Ferring Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No